CLINICAL TRIAL: NCT04839952
Title: Pilot Evaluation of a Healthy Lifestyle Intervention for Adolescent and Young Adult Survivors of Pediatric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00238848
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Cancer
Keywords: Pediatric cancer; Survivorship; Child; Adolescent; Weight; Obesity; Physical activity; Motivational interviewing; Problem solving; Culture; Exercise; Nutrition
MeSH Terms: conditions — Neoplasms; Body Weight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a small feasibility study. We will enroll 24 participants on the intervention arm and 12 participants to an education-only control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Lifestyles Intervention Arm (Experimental): Participants will receive the healthy lifestyles intervention.
  Interventions: Behavioral: Healthy Lifestyles
- Education-Only Control Arm (Active Comparator): Participants will receive the education-only intervention.
  Interventions: Behavioral: Education-Only Control

INTERVENTIONS:
Behavioral: Healthy Lifestyles — 12 telehealth sessions. The first 5 visits include psycho/medical education plus a motivational interviewing component. The second 7 sessions include psycho/medical education plus a problem solving training component.
  Arms: Healthy Lifestyles Intervention Arm
Behavioral: Education-Only Control — This control condition includes meeting with a clinician for one telehealth visit to review nutrition and physical activity recommendations.
  Arms: Education-Only Control Arm

SUMMARY:
This is a feasibility and acceptability trial to test a newly developed healthy lifestyle intervention for adolescent and young adult survivors of pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adolescents and young adults (15-25 years of age) who have completed cancer treatment at Johns Hopkins All Children's Hospital any time in the last five years. This age range was chosen because it corresponds to the recommended age range for cancer-related adolescents and young adult studies38.
* If the adolescent or young adult patient lives with a parent, other adult family member, or adult romantic/platonic partner, that person will also be invited to participate in the intervention as a support to the patient.
* If the adolescent or young adult patient lives with a parent or romantic partner, the parent or romantic partner will also be invited to participate in the intervention as a support to the patient. A parent or romantic partner is eligible to participate if the patient lives with them at least 50% of the time. The parent or romantic partner will not receive separate financial compensation for participation. Herein, we use the word "parent" only because we expect the vast majority of patients will live with a parent instead of a romantic partner. Patients who do not live with a parent or romantic partner will participate alone.
* The patient's cancer treatment must have included chemotherapy and/or radiation.
* If a patient's cancer relapses during the study period, the patient's oncologist must agree to the patient continuing in this intervention.

Exclusion Criteria:

* Potential participants who appear to have cognitive, motor, or language delays, as observed by research personnel or documented in the medical record, will be excluded from this study if delays preclude informed consent and/or study completion. Participants may request that research personnel read all assessment, education, and intervention materials aloud in a structured interview format, in which case participants could respond to items verbally and/or by pointing to visual aids. Because of this option, participants' ability to read and write are not requirements for participation.
* Because the motivational interviewing component of the intervention is language-dependent and requires significant time and training for certification in another language, non-English speaking patients will only be included in this study if the psychology postdoctoral fellow hired in this study is a native Spanish speaker and can demonstrate motivational interviewing proficiency in Spanish.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition knowledge as assessed by the General Nutrition Knowledge Questionnaire | Pre-intervention and 2 months after the intervention concludes
  Knowledge of nutrition recommendations, as evidenced by scores on the General Nutrition Knowledge Questionnaire - Revised (higher scores indicate greater knowledge).
Change in Physical activity knowledge as assessed by the Knowledge of American Heart Association Physical Activity Recommendations Questionnaire | Pre-intervention and 2 months after the intervention concludes
  Knowledge of physical activity recommendations, as evidenced by scores on the Knowledge of American Heart Association Physical Activity Recommendations Questionnaire (higher scores indicate greater knowledge).
Change in Physical activity as assessed by Fitbit data | Pre-intervention and 2 months after the intervention concludes
  Physical activity total weekly minutes, as evidenced by weekly Fitbit data (activity measured in minutes).
Change in Nutrition as assessed by the Rapid Eating Assessment for Patients score | Pre-intervention and 2 months after the intervention concludes
  Adherence to United States Department of Agriculture recommendations, as evidenced by the Rapid Eating Assessment for Patients (higher scores indicate better adherence to recommendations).
Intervention feasibility as assessed by the fidelity rating | Immediately following intervention
  Feasibility of conducting the intervention with high clinician fidelity, as evidenced by fidelity ratings for each session (fidelity represented as a percentage based on the extent to which the clinician covered all planned information for each session). Average intervention fidelity ratings should meet or exceed 80% fidelity.
Intervention acceptability as assessed by the Abbreviated Acceptability Rating Profile | Immediately following intervention
  Patient and caregiver acceptability of the newly developed intervention, as evidenced by the Abbreviated Acceptability Rating Profile (higher scores indicate greater acceptability, with scores equal to or greater than 30 indicating good acceptability per published standards).

SECONDARY OUTCOMES:
Change in Healthy lifestyle self-efficacy as assessed by the Weight Efficacy Lifestyle Questionnaire Short Form | Pre-intervention and 2 months after the intervention concludes
  Self-efficacy managing weight, as evidenced on scores on the Weight Efficacy Lifestyle Questionnaire Short Form (greater scores indicate greater self-efficacy).
Change in Healthy lifestyle self-efficacy as assessed by the Healthy Promoting Lifestyle Profile II | Pre-intervention and 2 months after the intervention concludes
  Self-efficacy maintaining healthy lifestyle behaviors, as evidenced by scores on the Healthy Promoting Lifestyle Profile II ((greater scores indicate greater self-efficacy).
Change in Body satisfaction as assessed by the Body Esteem Scale for Adults and Adolescents | Pre-intervention and 2 months after the intervention concludes
  Body satisfaction, as evidenced by scores on the Body Esteem Scale for Adults and Adolescents (higher scores indicate greater body satisfaction).
Change in Depression as assessed by the PROMIS Depressive Symptoms-Short Form | Pre-intervention and 2 months after the intervention concludes
  Depressive symptoms, as evidenced by scores on the PROMIS Pediatric Depressive Symptoms-Short Form or PROMIS Adult Depressive Symptoms-Short Form (greater scores indicate greater depressive symptoms).
Change in Anxiety as assessed by the PROMIS Anxiety Symptoms- Short Form | Pre-intervention and 2 months after the intervention concludes
  PROMIS Pediatric Anxiety Symptoms- Short Form or PROMIS Adult Anxiety Symptoms Short Form (greater scores indicate greater anxiety symptoms).
Change in Self-esteem as assessed by the Rosenberg Self Esteem Scale | Pre-intervention and 2 months after the intervention concludes
  Self-esteem, as evidenced by scores on the Rosenberg Self Esteem Scale (greater scores indicate greater self-esteem).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Faith, Ph.D., ABPP, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided